CLINICAL TRIAL: NCT07247370
Title: An Open-label Pilot Evaluation of Ketamine-Enhanced Psychotherapy in Individuals With Alcohol Use Disorder (AUD) and Co-morbid Major Depressive Disorder (MDD)
Brief Title: Ketamine-Enhanced Therapy for Individuals With Alcohol Use Disorder and Depression: A Pilot Study (KET-DUAL)
Acronym: KET-DUAL
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: South West Sydney Local Health District (Other)
Collaborators: The University of Sydney, Sydney, Australia (Unknown)
Responsible Party: Principal Investigator, Kirsten Morley BPsych MPH PhD, Professor, South West Sydney Local Health District
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X25-0138
Record Dates: First submitted 2025-11-16; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder (AUD); Major Depressive Disorder (MDD); Comorbidities and Coexisting Conditions
Keywords: Ketamine-enhanced psychotherapy; Open-label; Single-arm; Ketamine; Concurrent Treatment of AUD and comorbid MDD; Alcohol Use Disorder (AUD); Major Depressive Disorder (MDD)
MeSH Terms: conditions — Alcoholism; Depressive Disorder, Major | interventions — Ketamine; Cognitive Behavioral Therapy; Psychotherapy

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm, pilot study assessing the safety, feasibility, and preliminary efficacy of ketamine-enhanced therapy (KET) for individuals with alcohol use disorder (AUD) and co-morbid major depressive disorder (MDD) Participants will receive 3 doses of sub-anaesthetic ketamine combined with structured psychotherapy over six weeks, followed by follow-up assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketamine-enhanced therapy (KET): sub-anesthetic ketamine plus structured psychotherapy (Experimental): 1. x CBT session (Week 1)
     Dose 1: 1x Sub-anaesthetic subcutaneous dose of racemic ketamine (initially 0.7mg/kg, up to a potential maximum of 1.2mg/kg, at the discretion of the principal investigator and permitted based on tolerability) (Week 2)
  2. x CBT sessions (Week 2 - 3)
  Dose 2: 1x Sub-anaesthetic subcutaneous dose of racemic ketamine (initially 0.7mg/kg, up to a potential maximum of 1.2mg/kg, at the discretion of the principal investigator and permitted based on tolerability (Week 4)
  2 x CBT sessions (Week 4 - 5)
  Dose 3: 1x Sub-anaesthetic subcutaneous dose of racemic ketamine (initially 0.7mg/kg, up to a potential maximum of 1.2mg/kg, at the discretion of the principal investigator and permitted based on tolerability (Week 6)
  1x CBT session (Week 6)
  Interventions: Drug: Ketamine; Behavioral: Cognitive Behavioural Therapy

INTERVENTIONS:
Drug: Ketamine — Subcutaneous administration of of Ketamine across 3 dosing sessions (at week 2, 4 and 6). Dosing adjustments are permitted based on tolerability, with a minimum dose of 0.7mg/kg and a potential maximum of 1.2 mg/kg, at the discretion of the principal investigator (previous studies have found efficacy at 0.8mg/kg for AUD).
Behavioral: Cognitive Behavioural Therapy — This study uses a manualized CBT program adapted for ketamine-assisted context. It integrates evidence-based CBT for substance use and depression with principles of psychedelic-assisted therapy, including "set and setting." considerations central to psychedelic-assisted therapy. The therapist manual includes guidance on psychological preparation, intention-setting, integration, and therapeutic framing of ketamine experiences. Participants receive six 90-minute sessions over six weeks, delivered by trained health professionals (e.g., psychologists, mental health nurses, social workers) with specific training in the adapted CBT protocol and psychedelic-assisted therapy. Sessions include:
  Preparation (Week 1): Review of alcohol use, treatment goals, and ketamine orientation.
  Integration (Weeks 2, 4, 6): Post-dose processing and linking experience to recovery goals occurring 24-48 hours post dose.
  Continued CBT (Weeks 3, 5): Coping strategies, goal setting, and relapse prevention.
  Other Names: CBT; Psychotherapy

SUMMARY:
To assess the safety, feasibility and preliminary efficacy of ketamine-enhanced therapy (KET) for alcohol use disorder (AUD) and comorbid major depressive disorder (MDD) in an open-label, single arm, pilot clinical trial.

DETAILED DESCRIPTION:
New strategies for the treatment of alcohol use disorder (AUD) and co-morbid major depressive disorder (MDD) are urgently required. This population represents a high-risk group that has largely been excluded from addiction-focused trials despite its clinical complexity and poor response to standard interventions.

Recent early phase studies have shown that ketamine-enhanced psychotherapy (KET) can reduce alcohol consumption, enhance motivation and alleviate depressive symptoms. Effects have been shown to be particularly pronounced among participants who also received motivational enhancement therapy, suggesting a synergistic effect between ketamine and psychotherapy.

Emerging evidence suggests that KET may be of promise for AUD, and has demonstrated a good safety profile and potential efficacy in alcohol dependence. However, no trials to date have specifically targeted AUD and co-morbid MDD.

This project will assess the clinical safety, feasibility and preliminary efficacy of KET in individuals with AUD and co-morbid MDD. The investigators hypothesise that KET will be safe and feasible to deliver in this population, and expect to observe preliminary improvements in alcohol consumption, depressive symptoms, and treatment engagement. The KET intervention is also anticipated to be well tolerated with high levels of session attendance and acceptable rates of adverse events.

The trial will utilise an open-label, single-arm, pilot clinical trial design. A sample of 20 individuals will receive 6 weeks of treatment including 6 manualized cognitive-behavioural therapy sessions and 3 dosing sessions with Ketamine administered at 2 week intervals (0.7mg/kg initially up).

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe AUD according to the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-V) criteria
2. Presence of current Major Depressive Disorder (MDD), according to the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-V) criteria
3. Expressed motivation to reduce or cease alcohol consumption.
4. Consumed at least 21 standard drinks per week or 2 HDD per week (≥5 standard drinks/day for men; ≥4 for women) in the month prior to screening
5. Age 18-70
6. Adequate cognition and English language skills to give valid consent and complete research interviews
7. Stable housing
8. Willingness to give written informed consent.
9. Willingness to comply with study procedures and attend scheduled visits.

Exclusion Criteria:

1. DSM-5 diagnosis of current or past psychotic disorder, bipolar I disorder, or substance-induced psychosis.
2. Current acute suicidality, defined as high risk by the Columbia Suicide Severity Rating Scale (C-SSRS) or clinical judgment or attempts in the past 6 months.
3. DSM-5 diagnosis of current or past moderate-to-severe ketamine or other dissociative drug use disorder.
4. Use of ketamine (prescribed or non-prescribed) in the previous 4 weeks.
5. Enrolment in another interventional clinical trial that may interfere with safety, data quality, or trial participation.
6. Pregnant or breastfeeding, or planning to become pregnant during the course of the study.
7. Significant uncontrolled medical conditions, including but not limited to:

   * Severe or poorly controlled hypertension (>160/100 mmHg)
   * Severe cardiovascular disease (e.g., heart failure, recent myocardial infarction, dysrhythmia)
   * History of stroke, cerebral trauma, or intracranial mass/haemorrhage
   * Severe hepatic impairment (e.g., MELD ≥10) or end-stage liver disease, bladder or kidney disease
8. Clinically significant alcohol withdrawal at screening (e.g., CIWA-Ar ≥10, history of delirium tremens).
9. History of heightened intracranial pressure, seizures, or diagnosed seizure disorder (except childhood febrile seizures).
10. Known hypersensitivity to ketamine or any excipients.
11. Concurrent use of psychotropic medications (other than stable-dose antidepressants ≥4 weeks).
12. Active substance use disorder (moderate or severe) other than nicotine or caffeine; stable opioid use disorder permitted if on maintenance therapy (with strict stability criteria).
13. Inability or unwillingness to comply with study procedures, judged by the principal investigator.
14. Any clinically significant medical or psychiatric condition that, in the judgment of the Principal Investigator, poses a safety risk or could confound study results or hinder protocol adherence.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-04-10 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility will be assessed through recruitment rates, retention to follow-up, session attendance, and treatment adherence. | 22 weeks
  Feasibility outcomes will be assessed by the traffic light framework may be applied to guide progression decisions for future trials for each of the following variables: (i) time taken to recruit the sample; (ii) proportion of ineligible participants at (a) pre tele-screening and (b) onsite screening; (iii) number of participants who receive (a) at least two doses of ketamine and (b) at least four CBT sessions; (iv) retention rate over the trial. As this is the first study of its kind in this population and pilot studies are not generalisable to other contexts, these will be assessed and reported descriptively. Results will be synthesised in consideration of the feasibility to progress to larger studies, taking into account the measures described above. Specifically, based on our prior trials of CBT, pharmaco-assisted therapy and complex S9 trials, the following would be an estimation of failure to progress to full trial for each variable and when taken together: (i) > 24 months; (ii)
Safety will be assessed through the frequency, severity, and relatedness of adverse events (AEs), including dissociation, affective destabilisation, and vital sign abnormalities. | 22 weeks
  Safety outcomes including adverse events (AEs), serious adverse events (SAEs), and vital sign abnormalities, will be summarised descriptively across the study period. Feasibility outcomes (e.g., recruitment and retention rates, session attendance) will be analysed using proportions with corresponding 95% confidence intervals.

SECONDARY OUTCOMES:
Number of Heavy Drinking Days per week (HDDs) (>5 standard drinks/day for men; >4 for women) and total alcohol consumption. | 22 weeks
  This will be measured by the Timeline Follow Back and corroborated with Phosphatidylethanol (PEth) levels
Change in depressive symptoms measured by MADRS and DASS-21. | 22 weeks
  MADRS is a clinician-administered rating scale designed to assess the severity of depressive episodes in patients with mood disorders. It is widely used in clinical trials and psychiatric evaluations due to its sensitivity to treatment-related changes. The MADRS will be administered by trained health care professionals.
  The MADRS total score is calculated by summing the scores of 10 individual items, each rated on a scale from 0 to 6, yielding a total score range of 0 to 60. Higher scores indicate greater severity of depressive symptoms.
  The 10 items assessed in the MADRS include:
  Apparent sadness Reported sadness Inner tension Reduced sleep Reduced appetite Concentration difficulties Lassitude/Sluggishness Inability to feel (emotional capacity) Pessimistic thoughts Suicidal thoughts
  Each item is rated based on clinical judgment following a semi-structured interview, focusing on the past week.
  Clinically meaningful changes will be reported descriptively, including rates of ≥50%
Changes in suicidal ideation (weekly monitoring) using the Columbia Suicide Severity Rating Scale (C-SSRS). | 22 weeks
  The C-SSRS is a structured clinician-administered instrument with strong predictive validity for suicidal behavior, used in clinical and research settings to assess the presence, severity, and intensity of suicidal ideation and behavior. The C-SSRS is administered by trained clinicians.
  C-SSRS scoring includes four subscales: ideation severity (items 1-5, scored by the most severe type endorsed); intensity of ideation (sum of five items including frequency, duration, controllability, deterrents, and reasons for ideation; range 2-25; higher number indicates more intense ideation); suicidal behavior (presence or absence of actual, interrupted, aborted, or preparatory behavior recorded separately); and potential lethality (medical damage rated 0-5, potential lethality rated 0-2). At baseline, this is measured by the baseline version. At each visit following this, this will be recorded on the since last visit. Higher scores indicate more severe suicidality.
Changes in Positive and Negative Mood States | Week 2 (integration session 1), Week 4 (integration session 2), Week 6 (optional - at ketamine dose 3), Week 6 (integration session 3 and end of treatment)
  Mood states before/after ketamine sessions assessed by PANAS (Positive and Negative Affect Schedule). This will be measured at integration session 1 (week 2), 2 (week 4) and 3 (week 6). Used to measure an individual's emotional state, assessing two dimensions: Positive Affect (PA; captures feelings like enthusiasm and alertness), and Negative Affect (NA; measures distress and negative emotions like anger and anxiety).

OTHER OUTCOMES:
Changes in Depression | 22 weeks
  Measured by cumulative scores on the DASS-21 Depression Scale. This scale has a minimum score of 0 and maximum score of 21. A higher score indicates greater depression.
Changes in Anxiety | 22 weeks
  Measured by cumulative scores on the DASS-21 Anxiety Scale. This scale has a minimum score of 0 and maximum score of 21. A higher score indicates more anxiety.
Changes in Stress | 22 weeks
  Measured by cumulative scores on the DASS-21 Stress Scale. This scale has a minimum score of 0 and maximum score of 21. A higher score indicates more stress.
Change in Alcohol dependence severity | 22 weeks
  Measured by the Alcohol Dependence Scale. The minimum score is 0 and the maximum score is 47. A higher score indicates more severe dependence.
Sleep Quality | 22 weeks
  As measured by the PSQI (Pittsburgh Sleep Quality Index). This Index has a minimum score of 0 and a maximum score of 21. The higher the score indicates worse sleep quality.
Executive function, cognitive flexibility and task switching | 22 weeks
  To assess whether ketamine treatment improves executive functioning, specifically cognitive flexibility and task-switching ability, as measured by the Number-Letter Task (NLT). Key outcome measures include reaction time, accuracy, and switch cost (the performance difference between switch and repeat trials). Lower switch costs and faster, more accurate responses indicate improved executive control.
Executive functioning and cognitive flexibility | 22 weeks
  To assess whether ketamine treatment improves executive functioning and set-shifting, the Wisconsin Card Sorting Test (WCST) will be used.
  Participants are required to match stimulus cards based on varying classification principles (e.g., color, shape, number), which change without warning. Key outcome measures include the number of categories completed, total errors, perseverative responses, and perseverative errors. Higher performance is indicated by more categories completed and fewer perseverative errors, reflecting improved cognitive flexibility and executive control.
Changes in Alcohol Urge | 22 weeks
  To assess short term alcohol urge the Alcohol Urge Questionnaire (AUQ) will be used. This is a brief 8-item self-report questionnaire that evaluates acute alcohol craving as a single factor (unidimensional). Each item is rated on a Likert scale of 7 points, with higher scores indicating stronger urges to consume alcohol. Two of the questions are reversed scored.
Psychological inflexibility | 22 weeks
  As measured by the 7-item self-report Acceptance and Action Questionnaire, version 2 (AAQ-II). The items are rated on a 7-point Likert scale from 1 ("Never true") to 7 ("Always true"). Higher total scores are indicative of greater psychological inflexibility, while lower scores suggest more psychological flexibility. Scores between 24 and 28 are often used as a potential clinical cutoff indicating psychological distress.
Severity of pain and impact on functioning | 22 weeks
  Measured by The Brief Pain Inventory (BPI). Patients rate their current symptons, average experiences of pain and minimum and maximum intensities of symptoms on scales between 0 to 10. A total pain severity score can be found by averaging these individual items. Higher scores indicate greater severity and more interference. A score relating to impact on daily life can be calculated by averaging scores on each of the seven items, which also use scales from 0 to 10. Takes five minutes or less.
Withdrawal Status | At screening and prior to dosing (22 weeks).
  To determine changes in the severity of alcohol withdrawal symptoms the Revised Clinical Institute Withdrawal Assessment for Alcohol scale (CIWA-Ar) will be used. This 10-item scale evaluates common withdrawal symptoms including nausea/vomiting, tremor, paroxysmal sweats, anxiety, agitation, tactile disturbances, auditory disturbances, visual disturbances, headache and orientation. Each item is rated on a scale from 0 to 7 (except orientation, which is rated 0-4), with a total score ranging from 0 to 67. Higher scores indicate more severe withdrawal symptoms.
Drinking Diary | 22 weeks
  Daily texts will be sent out to participants querying the amount of alcohol they have consumed. Participant responses to this will be recorded. This will be managed through SEMA software.
Changes in Quality of Life | 22 weeks
  To assess whether treatment can improve quality of life as measured by the World Health Organization Quality of Life (WHOQOL-BREF). This 26-item questionnaire evaluates four domains of quality of life: physical health, psychological health, social relationships, and environment. Each item is rated on a 5-point Likert scale, and domain scores are transformed to a 0-100 scale. Higher scores indicate a better quality of life.
Treatment Satisfaction as measured by the CSQ-8 (client satisfaction questionnaire). | Week 1 (baseline) and week 10
  This instrument measures clients satisfaction with treatment. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Measurement of Drug Effect as measured by the PIQ-23 | PIQ will be completed on the day of an integration session at 2, 4 and 6 weeks.
  To assess whether treatment enhances acute psychologically insightful experiences we will use the Psychological Insight Questionnaire (PIQ-23).
  This 23-item self-report consists of two subscales: (a) Avoidance and Maladaptive Patterns Insights and (b) Goals and Adaptive Patterns Insights. The tool evaluates an individual's awareness and understanding of their own psychological processes, including recognition of patterns in thoughts, emotions, and behaviors. Each item is rated on a 5-point Likert scale, with higher scores indicating greater psychological insight.
CBT Session rating scale | 22 weeks
  As measured by the session rating scale (SRS). Following each CBT session, both the therapist and participant will complete a brief post-session rating. This scale measures; relationship, goals & topics, approach or method and overall psychotherapy session. Higher scores on each of these indicate a more positive experience.
Alcohol craving | 22 weeks
  As measured by the Penn Alcohol Craving Scale (PACS). 5-item self-report questionnaire that evaluates alcohol craving over the past week. Measures frequency, intensity, duration of craving, perceived control over drinking, and overall craving severity. Each item is rated on a 7-point Likert scale (0-6). Total scores range from 0 to 30, with higher scores indicating greater craving.
Cognitive function, specifically attention and executive control | Week 1 and week 10
  Assessed by the Stroop Task and Number-Letter Task at week 1 (baseline) and week 10.
Punishment insensitivity | Prior to MRI scan
  To assess whether ketamine treatment influences instrumental contingency learning and sensitivity to punishment, this will be measured by the Planets and Pirates Task. Key outcome measures include instrumental responses (e.g., click rates on each planet) and Pavlovian responses (e.g., active avoidance or shield use). Improved performance is indicated by increased avoidance of punished choices and enhanced detection of action-outcome contingencies.
Changes in Alcohol Craving | Before and after MRI scans at week 2, 4 and 6
  To assess whether ketamine treatment reduces acute alcohol craving across multiple dimensions, this will be measured by the Alcohol Craving Questionnaire Short Form-Revised (ACQ-SF-R). This 12-item questionnaire captures four factors: compulsivity, expectancy, purposefulness, and emotionality. Each item is rated on a Likert scale (strongly disagree - strongly agree), with higher scores indicating greater craving intensity. Takes less than 5 minutes to complete.
To measure changes in global cognitive functioning | Measured at screening and enrolment (visit 1, week 0), in addition to at follow-up 1 (visit 11, week 10)
  Global cognitive functioning assessed by the Montreal Cognitive Assessment (MoCA). The MoCA is a 30-point screening tool designed to detect mild cognitive impairment and assess multiple cognitive domains, including attention, concentration, executive functions, memory, language, visuospatial skills, conceptual thinking, calculations, and orientation. Higher scores indicate better cognitive performance, with a maximum score of 30.

CONTACTS AND LOCATIONS:
Locations (1):
- Drug Health Services, Royal Prince Alfred Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No